CLINICAL TRIAL: NCT04213872
Title: Gene Expression, Meditative Movement, and Emotional Distress (GME): A Pilot Study
Brief Title: Gene Expression, Meditative Movement, and Emotional Distress (GME)
Acronym: GME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: Children's Hospital Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GME Study (SITE00000289)
Record Dates: First submitted 2018-01-08; First posted 2019-12-30 (Actual); Results first posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-11

CONDITIONS: Cognitive Impairment
Keywords: breast cancer survivors; gene expression; emotional distress
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: This is a single-group nonrandomized pilot study on the effects of 8 weeks of MM program on changes in cognitive function, anxiety, sleep quality, depression, and selected gene expression factors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Meditative Movement (MM) (Experimental): The Meditative Movement (Qigong/Tai Chi Easy) program will be 8 weeks in duration with sessions once a week. Each session is approximately one hour. The PI will lead the MM sessions. The PI and the CRC will maintain contact with the MM group during the 8 weeks by telephone or in person.
  Interventions: Behavioral: Meditative Movement

INTERVENTIONS:
Behavioral: Meditative Movement — The Meditative Movement program is a blend of meditation and exercise based on Tai Chi and Qigong.

SUMMARY:
Study Title: Gene Expression, Meditative Movement and Emotional Distress (GME)

Background and Objectives:

Breast cancer survivors (BCS) often report decrements in cognitive functioning. Cognitive impairment (CI) is generally understood as resulting from chemotherapy or radiation, but may also result from chronic emotional distress experienced by breast cancer patients and survivors. Meditation and exercise are both known to reduce stress, with growing evidence for the potential of each to also improve cognitive functioning in cancer patients and survivors. A Meditative Movement (MM) program (Qigong/Tai Chi Easy) offers the potential of combining both benefits of meditation and exercise for breast cancer survivors. This is a pilot study, testing the MM program to effect changes in cognitive functioning and associated symptoms/conditions such as anxiety, depression, sleep quality and using gene expression factors as biomarkers to potentially measure the molecular signature of these changes. Forty BCS will be consented and assigned to an intensive eight week MM program. Cognitive functioning and associated symptoms/conditions will be assessed before and after the 8-week MM program to examine the participants' behaviors and symptoms. Peripheral blood samples will be collected before and after the 8-week MM program and will be analyzed for gene expression changes. If successful, this study may provide preliminary data for a full powered randomized control trial if results show promise in the psycho-behavioral outcomes and genomic expression results.

DETAILED DESCRIPTION:
This is a single-group pilot study on the effects of 8 weeks of MM practice on changes in cognitive function, anxiety, sleep quality, depression, and selected gene expression factors. Forty BCS will be consented and assigned to an intensive eight-week MM program. The forty BCS will be nonrandomly assigned to the eight-week MM program with no control group. The forty BCS will be organized in cohorts of 10 for the 8-week MM program. Cognitive functioning and associated symptoms/conditions data will be collected before and after the 8-week MM program to assess cognitive functioning, anxiety, depression, and sleep-quality. This data will be analyzed using the IBM SPSS Statistics program. Peripheral blood samples will be collected before and after the 8-week MM program. The gene expression data will be processed and analyzed by the bioinformatics team at the Single-Cell, Sequencing, and CyTOF Core (SC2), Children's Hospital Los Angeles (CHLA), Los Angeles.

Endpoints:

Endpoint 1: The Meditative Movement (MM) program will affect cognitive impairment.

Endpoint 2: The Meditative Movement (MM) program will affect anxiety, depression, and sleep quality.

Endpoint 3: The MM program will affect gene expression associated with cognitive impairment and associated symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Female patients diagnosed with breast cancer, Stage 0- III
* Between 6 months and 5 years past primary treatment
* 45 years of age and older
* Post-menopausal
* Speak or understand English

Exclusion Criteria:

* Women who are unable to stand (e.g., wheelchair or walker bound)
* Patients who are too weak or ill
* Women on antibiotics.
* Working night shift
* Anemia
* Uncontrolled diabetes

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Biologically Female
Enrollment: 27 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2020-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco V Munoz, Ph.D., Principal Investigator — Arizona State University
Locations (1):
- Robert and Beverly Lewis Family Cancer Care Center, Pomona, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Meditative Movement (MM) Group: minimum 45 years of age; female patients diagnosed with breast cancer, stages 0-III; between six months and five years past primary treatment; ability to speak or understand English; and post-menopausal for at least one year. Exclusion criteria: Women who were unable to stand (e.g., wheelchair or walker bound); patients who were too weak or ill; patients on antibiotics; women working on night shift; and patients with anemia or uncontrolled diabetes. Pregnant women, mentally disabled persons, and prisoners were excluded.
Period: Overall Study
Arm/Group | Meditative Movement (MM) Group
Started | 27
Completed | 14
Not Completed | 13

BASELINE CHARACTERISTICS:
Arm/Group | Meditative Movement (MM)
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 14
(FACT-COG)-Perceived Cog Impairment [Mean (Standard Deviation); unit: units on a scale] | 25.4 (14.2)
FACT-COG: Perceived Cognitive Abilities [Mean (Standard Deviation); unit: units on a scale] | 16.0 (5.1)
FACT-COG: Perceived Impairments on Quality of Life [Mean (Standard Deviation); unit: units on a scale] | 3.7 (3.8)
FACT-COG: Comments from Others [Mean (Standard Deviation); unit: units on a scale] | 1.5 (2.1)
Wechsler Adult Intelligence Scale (WAIS-III) 3rdEdition-letter/number Seq [Mean (Standard Deviation); unit: units on a scale] | 10.7 (3.2)
Wechsler Adult Intelligence Scale (WAIS-III) 3rdEdition -Digit Span Forward and Backward [Mean (Standard Deviation); unit: units on a scale] | 19.2 (4.8)
Pittsburgh Sleep Quality Index (PSQI) [Mean (Standard Deviation); unit: units on a scale] | 1.5 (0.8)
Profile of Mood States Short Form - Anxiety (POMS-SF) [Mean (Standard Deviation); unit: units on a scale] | 9.2 (7.7)
Profile of Mood States Short Form - Depression (POMS-SF) [Mean (Standard Deviation); unit: units on a scale] | 4.1 (4.9)
Brain derived neurotrophic factor (BDNF) [Mean (Standard Deviation); unit: fold change] | 0.11 (0.9)
Nuclear Factor kappa B (NF-kB1) [Mean (Standard Deviation); unit: fold change] | 171.7 (25.4)
Tumor Protein 53 (TP53) [Mean (Standard Deviation); unit: fold change] | 12.3 (2.7)

OUTCOME MEASURES:

1. Primary Outcome: Perceived Cognitive Impairments (CogPCI)
Description: Perceived Cognitive Impairments (CogPCI) is a patient self-report and validated subscale of the Functional Assessment of Cancer Therapy-Cognitive Function (FACT-COG), 20 items. The range of values are 0-80 with lower scores signifying better outcomes.
Time Frame: Measures data on cognitive functioning were collected one week before and one week after the 8-week MM program. Paired Sample t-test of SPSS were used to analyze data and report p-values within four weeks of final post-MM data collection.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Meditative Movement (MM) Group
Number analyzed (Participants) | 14
units on a scale | 17.3 (10.5)
Statistical Analysis 1: Comparison: Meditative Movement (MM) Group; Measure Pre-MM mean (sd) Post-MM mean (sd) Pre/Post MM mean (sd) difference P-Value CogPCI 25.4 (14.2) 17.3 (10.5) *-8.1 (3.7) .01 *reduction in scores indicate improvement; Test type: Other; p = .01, t-test, 2 sided

2. Primary Outcome: Perceived Cognitive Abilities (CogPCA)
Description: Perceived Cognitive Abilities (CogPCA) is a patient self-report and validated subscale of the Functional Assessment of Cancer Therapy-Cognitive Function (FACT-COG), 9 items. The range of values are 0-36 with higher scores signifying better outcomes.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Meditative Movement (MM): minimum 45 years of age; female patients diagnosed with breast cancer, stages 0-III; between six months and five years past primary treatment; ability to speak or understand English; and post-menopausal for at least one year. Exclusion criteria: Women who were unable to stand (e.g., wheelchair or walker bound); patients who were too weak or ill; patients on antibiotics; women working on night shift; and patients with anemia or uncontrolled diabetes. Pregnant women, mentally disabled persons, and prisoners were excluded.
Arm/Group | Meditative Movement (MM)
Number analyzed (Participants) | 14
units on a scale | 19.2 (5.3)
Statistical Analysis 1: Comparison: Meditative Movement (MM); Measure Pre-MM mean (sd) Post-MM mean (sd) Pre/Post MM mean (sd) difference P-Value CogPCA 16.0 (5.1) 19.2 (5.3) 3.2 (0.2) .03; Test type: Other; p = .03, t-test, 2 sided

3. Primary Outcome: Impact on Quality of Life (CogQOL)
Description: Impact on Quality of Life (CogQOL) is a patient self-report and validated subscale of the Functional Assessment of Cancer Therapy-Cognitive Function (FACT-COG), 4 items. The range of values are 0-16 with lower scores signifying better outcomes.
Time Frame: Measures data on associated symptoms/conditions were collected one week before and one week after the 8-week MM program. Paired Sample t-test of SPSS were used to analyze data and report p-values within four weeks of final post-MM data collection.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Meditative Movement (MM) Group
Number analyzed (Participants) | 14
units on a scale | 1.8 (2.2)
Statistical Analysis 1: Comparison: Meditative Movement (MM) Group; Measure Pre-MM mean (sd) Post-MM mean (sd) Pre/Post MM mean (sd) difference P-Value CogQOL 3.7 (3.8) 1.8 (2.2) *-1.9 (1.6) .04 *lower scores signifying better outcomes; Test type: Other; p = .04, t-test, 2 sided

4. Primary Outcome: Comments From Others (CogOth)
Description: Comments from Others (CogOth) is a patient self-report and validated subscale of the Functional Assessment of Cancer Therapy-Cognitive Function (FACT-COG), 4 items. The range of values are 0-16 with lower scores signifying better outcomes.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Meditative Movement (MM) Group
Number analyzed (Participants) | 14
units on a scale | 0.2 (0.4)
Statistical Analysis 1: Comparison: Meditative Movement (MM) Group; Measure Pre-MM mean (sd) Post-MM mean (sd) Pre/Post MM mean (sd) difference P-Value CogOth 1.5 (2.1) 0.2 (0.4) *-1.3 (1.7) .04 *lower scores signifying better outcomes; Test type: Other; p = .04, t-test, 2 sided

5. Primary Outcome: Wechsler Adult Intelligence Scale-Third Edition (WAIS-III): Letter-Number Sequencing
Description: WAIS-III: Letter-Number Sequencing measures working memory using letters and numbers in sequence recall. The scoring range is 0 to 21 with higher scores meaning better outcomes.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Meditative Movement (MM) Group
Number analyzed (Participants) | 14
units on a scale | 12.7 (2.8)
Statistical Analysis 1: Comparison: Meditative Movement (MM) Group; Measure Pre-MM mean (sd) Post-MM mean (sd) Pre/Post MM mean (sd) difference P-Value WAIS-III Letter/Number 10.7 (3.2) 12.7 (2.8) 2.0 (0.4) .01; Test type: Other; p = .01, t-test, 2 sided

6. Primary Outcome: Wechsler Adult Intelligence Scale-Third Edition (WAIS-III): Digit Span Forward and Backward
Description: WAIS-III): Digit Span Forward and Backward measures working memory using numbers in a series recall. The scoring range is 0 to 30 with higher scores meaning better outcomes.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Meditative Movement (MM) Group
Number analyzed (Participants) | 14
units on a scale | 19.7 (4.4)
Statistical Analysis 1: Comparison: Meditative Movement (MM) Group; Measure Pre-MM mean (sd) Post-MM mean (sd) Pre/Post MM mean (sd) difference P-Value WAIS-III Digit Span Forward and Backward 19.2 (4.8) 19.7 (4.4) 0.5 (0.4) .60; Test type: Other; p = .60, t-test, 2 sided

7. Primary Outcome: Pittsburg Sleep Quality Index (PSQI)
Description: The PSQI is a 19-item self-report questionnaire designed to assess sleep quality and disturbances over a I-month interval. The Pittsburgh Sleep Quality Index (PSQI): 19 items assess sleep, including subscales for subjective sleep quality, sleep latency, sleep duration, sleep disturbance, habitual sleep efficiency, daytime dysfunction and use of sleep medications. A global PSQI score >5 distinguishes good from poor sleepers. Lower scores mean better outcomes.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Meditative Movement (MM) Group
Number analyzed (Participants) | 14
units on a scale | 0.9 (0.7)
Statistical Analysis 1: Comparison: Meditative Movement (MM) Group; Measure Pre-MM mean (sd) Post-MM mean (sd) Pre/Post MM mean (sd) difference P-Value PSQI 1.5 (0.8) 0.9 (0.7) *-0.6 (0.1) .03 *Lower scores mean better outcomes; Test type: Other; p = .03, t-test, 2 sided

8. Primary Outcome: Profile of Mood States Short Form (POMS-SF) - Anxiety
Description: The POMs-SF consists of 37 items, adjectives scored on a 5-point Likert scale. POMS consists of the Total Mood Disturbance (TMD) dimensions (tension-anxiety; depression-dejection; anger-hostility; confusion-bewilderment. This pilot study reported results for the tension-anxiety TMD dimensions (12 items). Lower scores mean better outcomes.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Meditative Movement (MM) Group
Number analyzed (Participants) | 14
units on a scale | 4.2 (3.7)
Statistical Analysis 1: Comparison: Meditative Movement (MM) Group; Measure Pre-MM mean (sd) Post-MM mean (sd) Pre/Post MM mean (sd) difference P-Value POMS Anxiety 9.2 (7.7) 4.2 (3.7) *-5.0 (4.0) .05 *Lower scores mean better outcomes; Test type: Other; p = .05, t-test, 2 sided

9. Primary Outcome: Profile of Mood States Short Form (POMS-SF) - Depression
Description: The POMs-SF consists of 37 items, adjectives scored on a 5-point Likert scale. POMS consists of the Total Mood Disturbance (TMD) dimensions (tension-anxiety; depression-dejection; anger-hostility; confusion-bewilderment. This pilot study reported results for the depression-dejection TMD dimension (12 items). Lower scores mean better outcomes.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Meditative Movement (MM) Group
Number analyzed (Participants) | 14
units on a scale | 2.0 (3.0)
Statistical Analysis 1: Comparison: Meditative Movement (MM) Group; Measure Pre-MM mean (sd) Post-MM mean (sd) Pre/Post MM mean (sd) difference P-Value POMS Depression 4.1 (4.9) 2.0 (3.0) *-2.1 (1.9) .08 *Lower scores mean better outcomes; Test type: Other; p = .08, t-test, 2 sided

10. Secondary Outcome: Brain Derived Neurotropic Factor (BDNF) Gene Expression
Description: The BDNF gene regulates synaptic plasticity associated with cognitive functioning. Increased levels of BDNF gene expression are associated with improved cognitive functioning. Blood samples were collected post-intervention for RNA Sequencing to measure RNA levels as indicators of gene expression. Higher scores mean better outcomes.
Time Frame: Measures data on gene expression were collected one week before and one week after the 8-week MM program. Paired Sample t-test of SPSS were used to analyze data and report p-values within four weeks of final post-MM data collection.
Measure: Mean (Standard Deviation); unit: fold change
Arm/Group | Meditative Movement (MM)
Number analyzed (Participants) | 14
fold change | 0.30 (0.7)
Statistical Analysis 1: Comparison: Meditative Movement (MM); Measure Pre-MM mean (sd) Post-MM mean (sd) Pre/Post MM mean (sd) difference P-Value BDNF 0.11 (0.9) 0.30 (0.7) 0.19 (0.2) .30 Higher scores mean better outcomes; Test type: Other; p = .30, t-test, 2 sided

11. Secondary Outcome: Nuclear Factor Kappa B (NF-kB1) Gene Expression
Description: Decreased levels of NF-kB1 gene expression are associated with improvements in managing chronic stress. Blood samples were collected post-intervention for RNA Sequencing to measure RNA levels as indicators of gene expression. Lower scores indicate better outcomes.
Time Frame: as for outcome 10
Measure: Mean (Standard Deviation); unit: fold change
Arm/Group | Meditative Movement (MM)
Number analyzed (Participants) | 14
fold change | 173.7 (21.6)
Statistical Analysis 1: Comparison: Meditative Movement (MM); Measure Pre-MM mean (sd) Post-MM mean (sd) Pre/Post MM mean (sd) difference P-Value NF-kB1 171.7 (25.4) 173.7 (21.6) 2.0 (3.8) .80 Higher scores mean better outcomes; Test type: Other; p = .80, t-test, 2 sided

12. Secondary Outcome: Tumor Protein 53 (TP53) Gene Expression
Description: Increased TP53 gene expression is associated with suppressing cancer growth. Blood samples were collected post-intervention for RNA Sequencing to measure RNA levels as indicators of gene expression. Higher scores mean better outcomes.
Time Frame: as for outcome 10
Measure: Mean (Standard Deviation); unit: fold change
Arm/Group | Meditative Movement (MM)
Number analyzed (Participants) | 14
fold change | 13.1 (5.5)
Statistical Analysis 1: Comparison: Meditative Movement (MM); Measure Pre-MM mean (sd) Post-MM mean (sd) Pre/Post MM mean (sd) difference P-Value TP53 12.3 (2.7) 13.1 (5.5) 0.8 (2.8) .61; Test type: Other; p = .61, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 14 weeks
Description: In the context of this study, an adverse event is when a participant withdraws from the study due to physical or emotional discomfort. The PI or the Clinical Trials Coordinator (CRC) will report immediately any adverse events and monitoring results to the IRB coordinator.
Arm/Group | Meditative Movement (MM)
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

LIMITATIONS AND CAVEATS:
This study enrolled a small number of study participants, however, the results of this study parallel the results of larger studies conducted on the effects of meditation, exercise, and mind-body practices such as Yoga or Tai Chi/Qigong on the cognitive functioning, anxiety and quality of life factors for breast cancer survivors.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-13): https://cdn.clinicaltrials.gov/large-docs/72/NCT04213872/Prot_SAP_000.pdf